CLINICAL TRIAL: NCT04135274
Title: Is Neutrophil to Lymphocyte Ratio a Prognostic Factor of Sepsis in Newborns With Operated Neural Tube Defects?
Status: Completed | Type: Observational
Sponsor: Tepecik Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Firat Ergin, Medical Doctor, Tepecik Training and Research Hospital
Other Study IDs: 2018/12- 7
Record Dates: First submitted 2019-10-19; First posted 2019-10-22 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Neural Tube Defects; Newborn Sepsis
MeSH Terms: conditions — Neural Tube Defects; Neonatal Sepsis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sepsis group
  Interventions: Diagnostic Test: Neutrophil to lymphocyte ratio
- Non Sepsis group
  Interventions: Diagnostic Test: Neutrophil to lymphocyte ratio

INTERVENTIONS:
Diagnostic Test: Neutrophil to lymphocyte ratio — Neutrophil to lymphocyte ratio

SUMMARY:
We aimed to investigate whether Neutrophil Lymphocyte Ratio is a Prognostic Factor of Sepsis in Newborns with operated Neural Tube Defects?

ELIGIBILITY:
Inclusion Criteria:

* <28 days diagnosed with with neural Tüpe Defects To be operated

Exclusion Criteria:

* >28 days

Max Age: 28 Days | Sex: All
Age Groups: Child
Study Population: < 28 days infants
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Neutrophil to lymphocyte ratio is prognostic faktör for Sepsis | 3 years

IPD SHARING:
Plan to Share IPD: Undecided